CLINICAL TRIAL: NCT03082833
Title: Samsung Medical Center
Brief Title: Phase II Trial of AZD2014 in TSC1/2 Mutated or TSC1/2 Null GC Patients as Second-line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-016
Record Dates: First submitted 2017-02-16; First posted 2017-03-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD2014 50mg BD (Experimental): AZD2014 50mg BD continuous schedule of a 28 day cycle
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — AZD2014 is a selective dual mTOR kinase inhibitor targeting both mTORC1 (rapamycin sensitive) and mTORC2 (rapamycin insensitive) complexes of mammalian Target Of Rapamycin (mTOR).

SUMMARY:
Phase II trial of AZD2014 in TSC1/2 mutated or TSC1/2 null GC patients as second-line chemotherapy

DETAILED DESCRIPTION:
AZD2014 50mg BD continuous schedule of a 28 day cycle AZD2014 will be administered with orange juice in STG/TG patients. AZD2014 can be taken with or without food. The first dose of the day should be taken at approximately the same time each morning.The second dose of the day should be taken approximately 12 hours after the morning dose.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained doublet 5-fluoropyrimidine and platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as 1st line therapy.
   * Acceptable prior chemotherapy regimens for this protocol are chemotherapy regimens that include Immune Target agent therapy. (such as a pembrolizumab, ramucirumab etc)
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision of tumor sample (from eith tumor sample (from eith tumor sample (from eith tumor sample (from eith tumor sample (from eith er a resection or biopsy)er a resection or biopsy) er a resection or biopsy)er a resection or biopsy) er a resection or biopsy)er a resection or biopsy)er a resection or biopsy)er a resection or biopsy)er a resection or biopsy) er a resection or biopsy) er a resection or biopsy) er a resection or biopsy)er a resection or biopsy)
6. Patients with TSC1/2 mutation or null through the VIKTORY trial. (The VIKTORY trial uses Ion Torrent PGM to screen for a panel of cancer mutations and nanostring copy number variation panel (see addendum for the VIKTORY trial). Types of TSC1/2 mutation for this trial was defined in VIKTORY lab manual
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. ECOG performance status 0-2.
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

    - Haemoglobin ≥9.0 g/dL (transfusion allowed)
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * White blood cells (WBC) > 3 x 109/L
    * Platelet count ≥100 x 109/L (transfusion allowed)
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Serum creatinine ≤1.5 x institutional ULN
11. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
12. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.Or Patients must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: Post-menopausal - defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation

Exclusion Criteria:

* 1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.

  2. Any previous treatment with PIK3CA, AKT or mTOR inhibitor or agents with mixed PI3K / mTOR activity.

  3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.

  4. Patients unable to swallow orally administered medication. 5. Previous major surgery within 4 weeks prior to enrollment. 6. For AZD2014: Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment 8. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.

  9. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.

  10. Resting ECG with measurable QTcB > 450 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.

  11. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Left ventricular ejection fraction <55% measured by echocardiography, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment 12. Active or untreated brain metastases or spinal cord compression Patients with treated brain metastases or spinal cord compression are eligible if they have minimal neurologic symptoms, evidence of stable disease (for at least 1 month) or response on follow-up scan, and require no corticosteroid therapy for ≥ 1 week.

  13. Female patients who are breast-feeding or child-bearing 14. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV) 15. Patients with proteinuria (3+ on dipstick analysis )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | 6 months
  Objective response rate (ORR) by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea